CLINICAL TRIAL: NCT06659718
Title: Emulation of the Effects of Oral Semaglutide on Cardiovascular Outcomes in Individuals With Type 2 Diabetes and Established Atherosclerotic Cardiovascular Disease and/or Chronic Kidney Disease: SOUL Trial
Brief Title: Emulation of the SOUL Diabetes Trial in Healthcare Claims
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-SOUL
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral semaglutide: Exposure group
  Interventions: Drug: Oral semaglutide
- Sitagliptin: Reference group
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Oral semaglutide — New use of oral semaglutide dispensing claim is used as the exposure.
  Groups: Oral semaglutide
Drug: Sitagliptin — New initiation of sitagliptin dispensing claim is used as the reference.
  Groups: Sitagliptin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly emulated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not emulable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

The SOUL trial, which is a superiority trial to evaluate the effect of oral semaglutide versus placebo on MACE outcomes (CV death, nonfatal MI, or nonfatal stroke) among individuals with type 2 diabetes (T2DM) and established atherosclerotic cardiovascular disease (ASCVD) and/or chronic kidney disease (CKD).

The database study designed to emulate SOUL will be a new-user active comparative study, where we compare the effect of oral semaglutide versus sitagliptin on MACE outcome among patients with T2DM and with established ASCVD and/or CKD. Sitagliptin was selected to act as an active-comparator proxy for placebo.

Sitagliptin and the class of dipeptidyl peptidase-4 (DPP-4) inhibitors have been demonstrated not to have an effect on MACE in a series of RCTs, and they are used in similar stages of disease/line of therapy as semaglutide, as well as being similarly costly.

ELIGIBILITY:
Eligible cohort entry dates:

Market availability of oral semaglutide in the US began on 19th September 2019.

Optum: Study period between 20th Sept 2019 - 29th February 2024 Marketscan: Study period between 20th Sept 2019 - 31st Dec 2022 Medicare: Study period between 20th Sept 2019 - 31st Dec 2020

Inclusion Criteria:

* Type 2 diabetes mellitus
* Male or female, age equal to or above 50 years

At least one of the following conditions:

* Coronary heart disease defined by at least one of the following criteria:

  i. Prior myocardial infarction ii. Prior coronary revascularization procedure ii. 50% or above stenosis in coronary artery documented by cardiac catheterization, computerized tomography coronary angiography iv. Coronary heart disease with ischemia documented by stress test with any imaging modality
* Cerebrovascular disease defined by at least one of the following criteria:

  i. Prior stroke ii. Prior carotid artery revascularization procedure iii. 50% or above stenosis in carotid artery documented by x-ray angiography, magnetic resonance angiography, computerized tomography angiography or Doppler ultrasound
* Symptomatic peripheral artery disease (PAD) defined by at least one of the following criteria:

  i. Intermittent claudication with an Ankle-brachial index (ABI) below 0.85 at rest ii. Intermittent claudication with a 50% or above stenosis in peripheral artery (excluding carotid) documented by x-ray angiography, magnetic resonance angiography, computerized tomography angiography or Doppler ultrasound iii. Prior peripheral artery(excluding carotid) revascularization procedure iv. Lower extremity amputation at or above ankle due to atherosclerotic disease (excluding trauma or osteomyelitis)
* Chronic kidney disease defined as: i. eGFR below 60mL/min/1.73 m^2 (based on medical records using latest available and no more than 6 months old assessment)

Exclusion Criteria:

* Any of the following: myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischemic attack within the past 60 days prior to the day of screening
* Heart failure presently classified as being in New York Heart Association Class IV
* Treatment with any glucagon-like peptide-1 receptor agonist within 30 days before screening
* Semaglutide
* History of MEN-2 or family history of medullary thyroid cancer
* History of pancreatitis
* History of or planning bariatric surgery, including banding procedures or surgical gastric and/or intestinal bypass
* Plans for pregnancy during the course of the study for women of child-bearing potential
* History of cancer, other than non-melanoma skin cancer, that required therapy in the 5 years prior to randomization
* Chronic or intermittent hemodialysis or peritoneal dialysis or severe renal impairment (corresponding to eGFR <30 ml/min/1.73 m2)
* Proliferative retinopathy or maculopathy requiring acute treatment
* History of diabetic ketoacidosis
* Missing age or gender
* Nursing home admission

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population included patients aged 50 years or older with type 2 diabetes (T2DM) and established atherosclerotic cardiovascular disease (ASCVD) and/or chronic kidney disease (CKD).
Sampling Method: Non-Probability Sample
Enrollment: 43650 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE), including myocardial infarction, stroke and all cause death | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  Hazard ratio

OTHER OUTCOMES:
Cataract surgery (negative control) | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  Hazard ratio

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT06659718/Prot_SAP_003.pdf